CLINICAL TRIAL: NCT06564792
Title: CoMBo Study: Contingency Management for Both HIV And Stimulant Use in Primary Care
Brief Title: Contingency Management in HIV Care for Both Stimulant Use & ART Adherence
Acronym: CoMBo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-38747
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Stimulant Use (Diagnosis); Hiv
MeSH Terms: conditions — Disease; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contingency management arm (Experimental): Participants are offered once weekly contingency management in clinic to support reduced stimulant use and HIV medication adherence.
  Interventions: Behavioral: Contingency management

INTERVENTIONS:
Behavioral: Contingency management — Once weekly contingency management visit involving 15 minutes+ of motivational interviewing and provision of incentives for stimulant-negative urine tests and/or tenofovir-positive urine tests.

SUMMARY:
Methamphetamine use and associated sequelae have been rising, and represent a major barrier to successful control of the HIV epidemic. Methamphetamine use is associated with poor adherence to antiretroviral therapy for HIV, and the investigators propose a trial of contingency management (providing incentives for behavioral change) targeting both reduced methamphetamine use and improved adherence to HIV medications. The investigators will utilize a real-time, point-of-care urine assay for both outcomes, aiming to evaluate feasibility, acceptability and preliminary effectiveness of HIV care-based contingency management. Hair levels will also be studied as a quantitative outcome for reduction in methamphetamine use.

DETAILED DESCRIPTION:
Methamphetamine (MA) use is increasing in the United States, along with a sharp rise in overdose deaths. MA use is particularly prevalent among people with HIV (PWH), which can contribute to non-adherence to antiretroviral therapy (ART) and progression to AIDS. Contingency management (CM) is an evidence-based intervention that has repeatedly demonstrated efficacy in stimulant use disorder treatment and has also proved efficacious in improving ART adherence for those in care. Since uptake of CM outside of formal drug treatment programs has been limited, incorporating CM into HIV primary care is an important opportunity to expand access to treatment for MA use disorder while also supporting ART adherence.

This study addresses two barriers that have each limited outward expansion of CM into HIV primary care: 1) feasibility challenges for CM in clinical practice settings; as CM is traditionally delivered 2-3x weekly, this study explores a de-intensified CM schedule (e.g., once weekly visits) in HIV primary care; and 2) CM for ART adherence has been previously limited by the inaccuracy of indirect or non-timely measures of adherence.

The study utilizes a novel point-of-care urine tenofovir assay to perform POC testing on the same urine specimen for both ART use and MA non-use, enabling a truly paired CM intervention that addresses the following aims: 1) a pilot RCT evaluating feasibility of de-intensified (once weekly) combined contingency management for reducing MA use and increasing ART adherence in HIV primary care, compared to conventional twice weekly CM; 2) in-depth interviews following RCT completion to qualitatively explore the acceptability of this intervention to participants and their primary care providers; and 3) given incomplete ability to detect cumulative MA use with only once weekly urine testing, the investigators will study the correlation between monthly MA hair levels with monthly Timeline Followback interviews to validate use of hair MA levels to be able to quantitatively detect reduced use (in addition to abstinence) as a future study outcome.

ELIGIBILITY:
Inclusion Criteria:

* Stimulant use disorder
* Living with HIV or risk for HIV
* Suboptimal ART adherence (treatment or prevention)

Exclusion Criteria:

* Unable to provide urine testing weekly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility: proportion of CM visits attended | Measured during intervention participation.
  The investigators will report multiple process measures as feasibility outcomes, though primary outcome is the number and proportion of contingency management visits attended (of 12). It is expected that 50% of participants will attend at least 6 or more CM visits, which is defined as minimum engagement suggesting feasibility of this HIV primary care-based CM intervention.
Acceptability: in-depth interviews with participants, staff | Interviews performed within 6 months of intervention participation.
  The investigators will conduct in-depth qualitative interviews to understand factors and circumstances that influence CM engagement among PWH with stimulant use disorder and suboptimal ART adherence. These findings will also help elucidate mechanisms contributing to stimulant use reduction and ART adherence when once weekly CM is delivered to PWH in a designated primary care setting.

SECONDARY OUTCOMES:
Effectiveness (Urine) | Measured during intervention participation.
  The investigators will report proportion of urine tests negative for stimulants; proportion positive for tenofovir.
Effectiveness (Hair) | Analyzed within 1 year following hair collection
  The investigators will correlate within-person changes in cumulative stimulant hair levels with the days free of stimulant use performed pre- vs. post-intervention using mixed effects Poisson regression with random effects for individual.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Appa, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF at San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steiner G, Baral S, Riley ED, Shoptaw S, Chamie G, Roberts K, Suchman L, Knight K, Gandhi M, Coffin P, Appa A. Harm Reduction Contingency Management for Stimulant Use Reduction and Antiretroviral Therapy Adherence in HIV Primary Care: Protocol for an Implementation Effectiveness Study. JMIR Res Protoc. 2025 Aug 18;14:e67292. doi: 10.2196/67292. PMID 40825537